CLINICAL TRIAL: NCT05154695
Title: Precision Medicine for Sng/Pain Control
Acronym: SNG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202011007RIND
Record Dates: First submitted 2021-10-12; First posted 2021-12-13 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2022-12

CONDITIONS: Rehabilitation; Pain, Shoulder; Pain, Chronic
Keywords: sng/pain; Low-level Laser Therapy; ultrasound; prolotherapy; next generation sequencing
MeSH Terms: conditions — Shoulder Pain; Chronic Pain | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: The eligible participants first received LLLT with a 685-nm wavelength and an output of 30 mW at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle.
  They are randomly assigned into two groups (40 subjects in each group): A. therapeutic ultrasound group; B. prolotherapy group. The same physician (the principal investigator) injects all participants to avoid inter-physician variability. No other medication or physical modality was given to avoid efficacy interference in both groups.
  Rescue therapy (cross-over treatment): If the participant does not satisfy with their first round treatment and the improvement of VAS is less than 1.0, then they are eligible to receive the rescue therapy-the treatment in the other group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A.therapeutic ultrasound group (Active Comparator): Group A receives 1 MHz therapeutic ultrasound for 5 min at a frequency of 2-3 times per week at the painful upper trapezius muscle.
  Interventions: Device: LASER; Device: A.therapeutic ultrasound group; Drug: B.prolotherapy group
- B.prolotherapy group (Active Comparator): Group B receives hypertonic prolotherapy at perimysium of upper trapezius muscle. The injectant is 5ml 5% dextrose solution.
  Interventions: Device: LASER; Device: A.therapeutic ultrasound group; Drug: B.prolotherapy group

INTERVENTIONS:
Device: LASER — The eligible participants first received LLLT with a 685-nm wavelength and an output of 30 mW at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle.
Device: A.therapeutic ultrasound group — Group A receives 1 MHz therapeutic ultrasound for 5 min at a frequency of 2-3 times per week at the painful upper trapezius muscle.
  Other Names: Group A
Drug: B.prolotherapy group — Group B receives hypertonic prolotherapy at perimysium of upper trapezius muscle. The injectant is 5ml 5% dextrose solution.
  Other Names: Group B

SUMMARY:
Patients have different response to different treatment modalities, and sore/pain medicine is no exception. In our experience, low-level laser (LLL), ultrasound, and prolotherapy can reduce sore /pain through different genetic pathway. Whether the therapeutic effect is controlled by the genetic variants of those sore /pain related genes or not, is still in debate. The aims of this study are (1) To find genetic SNPs which can determine the response of sore /pain treatment modalities. (2) To find possible metabolomics and proteomic markers of sore /pain. (3) To determine the algorithm of precision medicine for sore /pain control via the genetic markers. Investigators will recruit 80 myofascial pain patients from Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital Bei-Hu Branch in 2021 and 2022. The participants will receive LLL, ultrasound, and prolotherapy, and the therapeutic effect will be recorded. The blood and urine samples from the first, the second, and the third visits will be analyzed by next generation sequencing, and mass spectrometry to find the possible biomarker in 2023 and 2024. Investigators expect to develop the individualized treatment plan by means of these biomarkers. Hopefully, the results will be widely applied in the field of sore /pain medicine.

DETAILED DESCRIPTION:
Pain is defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage or described in terms of such damage" by the International Association for the Study of Pain (IASP). The musculoskeletal disorders are not only the most common cause of chronic sore/pain, but they also result in significant disability in about 50% of sufferers in the US. Furthermore, since these disorders are the most common cause of severe, long-term pain and disability in the elderly over 65 years. In the practice of pain medicine, the doctors predominantly use multi-modal treatment, including medications, physical agents, and injection, to relieve patients' discomfort.

In the past years, our team had some achievements to justify the search of genetic variants for development of a new sore/pain treatment algorithm.

(1) Analgesia of LLLT is through TRPV1. (2) Analgesia by therapeutic ultrasound is through ASIC3. (3) Dextrose injection decreased chronic muscle pain through ASIC1a. (4) Biomarker for sore/pain in fibromyalgia.

According to the clinical outcome, some patients responded to physical agents well, and some preferred injections. The genetic variants of the above-mentioned genes might be the determining factors of differential therapeutic effects. However, it took about 4-8 weeks for a patient to switch from one treatment option to another one. If investigators can determine the optimal treatment modality by genetic biomarkers, the treatment course and total expanse will decrease a lot.

Investigators hypothesize that the genetic variants of the proposed genes (TRPV1, ASIC1a, ASIC3, Tac1, COMT, TCL1A, POMC, RGS4, ASIC2, ASIC4, TRPA1, NK1R, G2A, GPR4, OGR1, TDAG8, TASK1, TASK2, TASK3, TREK1, P2X2, P2X3, P2X5, TRPV4, KCNK1, NTSR1, NTSR2) could be the prognostic biomarkers of sore /pain treatments. Our specific Aims are:

1. To set up next generation sequencing (NGS)-based approach to find genetic variants which can determine the response of sore/pain treatment modalities.
2. To find possible metabolomics and proteomic markers of sore/pain.
3. To determine the algorithm of precision medicine for sore/pain control via the genetic markers.

Six. study design I Patient eligibility Investigators will recruit patients from National Taiwan University Hospital Bei-Hu Branch.

Inclusion criteria: (1) Age between 20-100 years old. (2) Diagnosed as myofascial pain syndrome patients and willing to receive treatment (including LLLT, therapeutic ultrasound, and local dextrose injection therapy). The diagnosis of MPS was confirmed by the Principal Investigator using the criteria of taut band, trigger point, and radiating pain.

Exclusion criteria: Those having active infection, malignancy, and hematological diseases were excluded. The patients had received local injection at upper trapezius within 3 months are also excluded.

II Study design and flow

1. After obtaining the informed consent, the basic demographic data, including age, gender, job, education level, and past medical history of eligible patients are collected.
2. The eligible patients first received LLLT with a 685-nm wavelength and an output of 30 mW at energy densities of 8 J/cm2 at trigger point of upper trapezius muscle. The pre- and post-treatment VAS-pain and VAS-sng are collected for LLLT phenotype determination, respectively.
3. Then, they are randomly assigned into two groups (40 subjects in each group): A. therapeutic ultrasound group; B. prolotherapy group. Group A receives 1 MHz therapeutic ultrasound for 5 min at a frequency of 2-3 times per week at the painful upper trapezius muscle. Group B receives hypertonic prolotherapy at perimysium of upper trapezius muscle. The injectant is 5ml 5% dextrose solution. To ensure that the needle was not in a blood vessel, the needle was aspirated before injection. The same physician (the principal investigator) injects all patients to avoid inter-physician variability. No other medication or physical modality was given to avoid efficacy interference in both groups.
4. The recruited patients receive evaluation before and after injection, and 2-week after injection. The primary outcome is VAS-pain and VAS-sore (visual analogue scale) with a score of 0-100, where 100 is the value representing the highest degree of pain. The secondary outcomes are pain threshold, muscle tone, and SF-36-a questionnaire consists of 36 items and 8 domains addressing the patient's perception of their QoL. Venous blood and urine samples were collected at first visit and 2-week visit, respectively. The blood samples were labeled with an anonymized ID number, centrifuged, and stored at -80 ºC in a locked freezer until the time of future processing. The buffy coat is separated after centrifugation, and stored as well. The urine samples were aliquoted and stored at -80 ºC in a locked freezer for future analysis.
5. Rescue therapy (cross-over treatment): If the participant does not satisfy with their first round treatment and the improvement of VAS is less than 1.0, then they are eligible to receive the rescue therapy-the treatment in the other group. And they will return to clinic for another 2 weeks. The outcome variables will be collected in the 3rd visit as well.

(1) DNA extraction and NGS-based sequencing and genotyping Genomic DNA will be extracted from peripheral blood mononuclear cells of the participants using the Gentra Puregene kit following the protocol from the manufacturer, and subjected to agarose gel and O.D. ratio tests to confirm its purity and concentration. DNA will be fragmented using Covaris, aiming at the peak length of 800 bp. Illumina libraries will be generated from gDNA using TruSeq Library Preparation Kit.

DNA capture probes will be custom-designed to target TRPV1, ASIC1a, ASIC3, Tac1, COMT, TCL1A, POMC, RGS4, ASIC2, ASIC4, TRPA1, NK1R, G2A, GPR4, OGR1, TDAG8, TASK1, TASK2, TASK3, TREK1, P2X2, P2X3, P2X5, TRPV4, KCNK1, NTSR1, NTSR2 and will be synthesized using the Roche KAPA HyperChoice protocol. All the coding regions and non-coding regions (promoters, introns, 5' and 3' untranslated regions) of these 8 genes will be included.

NGS target region enrichment will be applied to enrich/capture the target region (~148 Kb). The enriched libraries will then be sequenced using Illumina MiSeq to generate paired-end reads of 300 bp. The expected depth of the targeted regions will be 200x on average.

(2) Metabolomic and proteomic analysis

1. Briefly, The LC-MS analyses of urine and serum involved using an Agilent 1290 UPLC system (ACQUITY UPLC HSS T3 column, 2.1×100 mm; 1.8 µm; Waters, Milford, MA, USA) coupled with the 6540-Quadrupole-Time-of-Flight (QTOF) mass system (Agilent Technologies, Santa Clara, CA, USA). MS raw files were converted to the mzXML format using Trapper (ISB) and processed by TIPick, an in-house package. After TIPick processing, the scaling-based normalization was performed according to the total ion abundances from each UHPLC-MS data set.
2. The LC-MS lipidomic profiling was performed and described in detail. Concisely, lipidomic profiling was run on a ZORBAX Eclipse Plus C18 (2.1 x 100 mm, 1.8 µm, Agilent Technologies, Waldbronn, Germany) for QTOF, as well as mobile phase A consisted of 0.1% aqueous formic acid and 10 mM ammonium acetate and mobile phase B consisted of 0.1% formic acid and 10 mM ammonium acetate in ACN/isopropyl alcohol (50/50). The autosampler and column oven were maintained at 4°C and 55°C, respectively. The injection volume was 5 μl. MS acquisition was executed in the precursor ion scan (PIS) mode and multiple reaction monitoring (MRM) mode.
3. All UPLC-MS raw data were converted to mzXML format by using Trapper (ISB) and normalized by TIPick, an in-house package, as well as peak enhancement and peak chosen for the targeted metabolites. An in-house database of sphingomyelins (SM), lysophosphatidylcholine (LysoPC), ceramides (Cer), phosphatidylcholines (PCs), phosphatidylinositol (PI), phosphatidylethanolamine (PE), and cerebroside (CB) in the Metabolomics Core Laboratory, Center of Genomic Medicine, National Taiwan University, was used for screening.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age between 20-100 years old.
* (2) Diagnosed as myofascial pain syndrome patients and willing to receive treatment (including LLLT, therapeutic ultrasound, and local dextrose injection therapy).

Exclusion Criteria:

* Those having active infection, malignancy, and hematological diseases were excluded. The patients had received local injection at upper trapezius within 3 months are also excluded.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) - first | Baseline Visual Analogue Scale
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-10. score 0 means 'no pain' and score 10 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(1-4 point), moderate pain (5-7 point ), and severe pain (8-10 point).
Visual Analogue Scale (VAS) - second | Change from Baseline Visual Analogue Scale at 2 weeks.
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-10. score 0 means 'no pain' and score 10 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(1-4 point), moderate pain (5-7 point ), and severe pain (8-10 point).
Visual Analogue Scale (VAS) - third | Change from Baseline Visual Analogue Scale at 4 weeks (if crossover).
  Visual Analogue Scale (VAS) anchor the patient's mark, providing a range of scores from 0-10. score 0 means 'no pain' and score 10 means 'pain worst'. VAS have been recommended: no pain (0 point), mild pain(1-4 point), moderate pain (5-7 point ), and severe pain (8-10 point).

SECONDARY OUTCOMES:
SF-36 | Baseline, week 2, week 4 (if crossover)
  Quality of life (36-Item Short Form Survey)
Pain thresholds | Baseline, week 2, week 4 (if crossover)
  Pain thresholds range from 0 to 800. Low thresholds means higher pain sensitivity (Pain tolerance) or muscle inflammation.
Myoton-Muscle tone | Baseline, week 2, week 4 (if crossover)
  Muscle tone means state of muscle tension, which unit is Natural oscillation frequency [Hz]. This higher or lower value meaning is uncertainty. The range was from 10 to 30 Hz.
Myoton- Dynamic stiffness | Baseline, week 2, week 4 (if crossover)
  Muscle tone means muscle biomechanical properties, which unit is N/m. This higher or lower value meaning is uncertainty. The range was from 100 to 600 Hz.

CONTACTS AND LOCATIONS:
Overall Officials: Der-Sheng Han, Physician, Study Director — International Committee of Medical Journal Editors
Locations (1):
- National Taiwan University Hospital Bei-Hu Branch, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data doesn't shared with other researchers.

REFERENCES:
- [Background] Avrampou K, Pryce KD, Ramakrishnan A, Sakloth F, Gaspari S, Serafini RA, Mitsi V, Polizu C, Swartz C, Ligas B, Richards A, Shen L, Carr FB, Zachariou V. RGS4 Maintains Chronic Pain Symptoms in Rodent Models. J Neurosci. 2019 Oct 16;39(42):8291-8304. doi: 10.1523/JNEUROSCI.3154-18.2019. Epub 2019 Jul 15. PMID 31308097
- [Background] Chang KV, Wu WT, Han DS, Ozcakar L. Static and Dynamic Shoulder Imaging to Predict Initial Effectiveness and Recurrence After Ultrasound-Guided Subacromial Corticosteroid Injections. Arch Phys Med Rehabil. 2017 Oct;98(10):1984-1994. doi: 10.1016/j.apmr.2017.01.022. Epub 2017 Feb 27. PMID 28245972
- [Background] Collins FS, Varmus H. A new initiative on precision medicine. N Engl J Med. 2015 Feb 26;372(9):793-5. doi: 10.1056/NEJMp1500523. Epub 2015 Jan 30. PMID 25635347
- [Background] Genovese TJ, Mao JJ. Genetic Predictors of Response to Acupuncture for Aromatase Inhibitor-Associated Arthralgia Among Breast Cancer Survivors. Pain Med. 2019 Jan 1;20(1):191-194. doi: 10.1093/pm/pny067. PMID 29912452
- [Background] Hsu WH, Lee CH, Chao YM, Kuo CH, Ku WC, Chen CC, Lin YL. ASIC3-dependent metabolomics profiling of serum and urine in a mouse model of fibromyalgia. Sci Rep. 2019 Aug 20;9(1):12123. doi: 10.1038/s41598-019-48315-w. PMID 31431652
- [Background] Hsu WH, Wang SJ, Chao YM, Chen CJ, Wang YF, Fuh JL, Chen SP, Lin YL. Urine metabolomics signatures in reversible cerebral vasoconstriction syndrome. Cephalalgia. 2020 Jun;40(7):735-747. doi: 10.1177/0333102419897621. Epub 2020 Jan 7. PMID 31910660
- [Background] Li L, Wang HM, Shen Y. Chinese SF-36 Health Survey: translation, cultural adaptation, validation, and normalisation. J Epidemiol Community Health. 2003 Apr;57(4):259-63. doi: 10.1136/jech.57.4.259. PMID 12646540
- [Background] Liao HW, Kuo CH, Chao HC, Chen GY. Post-column infused internal standard assisted lipidomics profiling strategy and its application on phosphatidylcholine research. J Pharm Biomed Anal. 2020 Jan 30;178:112956. doi: 10.1016/j.jpba.2019.112956. Epub 2019 Oct 30. PMID 31704131
- [Background] Lin YH, Wu CC, Lin YH, Lu YC, Chen CS, Liu TC, Chen PL, Hsu CJ. Targeted Next-Generation Sequencing Facilitates Genetic Diagnosis and Provides Novel Pathogenetic Insights into Deafness with Enlarged Vestibular Aqueduct. J Mol Diagn. 2019 Jan;21(1):138-148. doi: 10.1016/j.jmoldx.2018.08.007. Epub 2018 Sep 28. PMID 30268946
- [Background] Loeser JD, Treede RD. The Kyoto protocol of IASP Basic Pain Terminology. Pain. 2008 Jul 31;137(3):473-477. doi: 10.1016/j.pain.2008.04.025. Epub 2008 Jun 25. No abstract available. PMID 18583048
- [Result] Cho CH, Lho YM, Ha E, Hwang I, Song KS, Min BW, Bae KC, Kim DH. Up-regulation of acid-sensing ion channels in the capsule of the joint in frozen shoulder. Bone Joint J. 2015 Jun;97-B(6):824-9. doi: 10.1302/0301-620X.97B6.35254. PMID 26033064
- [Result] Han DS, Lee CH, Shieh YD, Chen CC. Involvement of Substance P in the Analgesic Effect of Low-Level Laser Therapy in a Mouse Model of Chronic Widespread Muscle Pain. Pain Med. 2019 Oct 1;20(10):1963-1970. doi: 10.1093/pm/pnz056. PMID 30908578
- [Result] Hsiung YC, Lin PC, Chen CS, Tung YC, Yang WS, Chen PL, Su TC. Identification of a novel LDLR disease-causing variant using capture-based next-generation sequencing screening of familial hypercholesterolemia patients in Taiwan. Atherosclerosis. 2018 Oct;277:440-447. doi: 10.1016/j.atherosclerosis.2018.08.022. PMID 30270083
- [Result] Lin JH, Hung CH, Han DS, Chen ST, Lee CH, Sun WZ, Chen CC. Sensing acidosis: nociception or sngception? J Biomed Sci. 2018 Nov 29;25(1):85. doi: 10.1186/s12929-018-0486-5. PMID 30486810
- [Result] Niculescu AB, Le-Niculescu H, Levey DF, Roseberry K, Soe KC, Rogers J, Khan F, Jones T, Judd S, McCormick MA, Wessel AR, Williams A, Kurian SM, White FA. Towards precision medicine for pain: diagnostic biomarkers and repurposed drugs. Mol Psychiatry. 2019 Apr;24(4):501-522. doi: 10.1038/s41380-018-0345-5. Epub 2019 Feb 12. PMID 30755720
- [Result] Park G, Kim CW, Park SB, Kim MJ, Jang SH. Reliability and usefulness of the pressure pain threshold measurement in patients with myofascial pain. Ann Rehabil Med. 2011 Jun;35(3):412-7. doi: 10.5535/arm.2011.35.3.412. Epub 2011 Jun 30. PMID 22506152
- [Result] Rabago D, Yelland M, Patterson J, Zgierska A. Prolotherapy for chronic musculoskeletal pain. Am Fam Physician. 2011 Dec 1;84(11):1208-10. No abstract available. PMID 22150651